CLINICAL TRIAL: NCT03932955
Title: Study Evaluating the Efficacy and Safety of MC-19PD1 CAR-T in Relapsed or Refractory B Cell Lymphoma
Brief Title: MC-19PD1 CAR-T in Relapsed or Refractory B Cell Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Jun Zhu, Director, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC-19PD1 CART201902
Record Dates: First submitted 2019-04-22; First posted 2019-05-01 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MC-19PD1 CAR-T Cells (Experimental)
  Interventions: Biological: MC-19PD1 CAR-T cells

INTERVENTIONS:
Biological: MC-19PD1 CAR-T cells — T cells purified from the PBMC of subjects, transduced with anti-CD19 CAR and PD1/CD28 chimera lentiviral vector, expanded in vitro for future administration.

SUMMARY:
This is a single center, single arm, open-lable phase 1 study to determine the safety and efficacy of CD19-CAR-T cells in patients with relapsed or refractory B-cell lymphoma.

DETAILED DESCRIPTION:
In this single-center, open-label, nonrandomized, no control, prospective clinical trial, appoximately 15 relapsed or refractory B-cell lymphoma patients will be enrolled. Side effects of CD19 CAR T cells therapy will be monitored. The purpose of current study is to determine the clinical efficacy and safety of CD19 CAR T cells therapy in patients with R/R B-cell lymphoma

ELIGIBILITY:
Inclusion Criteria:

（1）CD19 positive B-cell lymphoma; （2）Relapsed and refractory B-cell lymphoma: patients previously received at least first-line and second- line treatment and fail to achieve CR; （3）At least 1 measurable tumor foci according to the 2014 Lugano treatment response criteria; （4）18 to 70 Years Old, Male and female; （5）Expected to survive for more than 3 months; （6）Clinical performance status of ECOG score 0-1; （7）Important organ function is satisfied: cardiac ultrasound indicates cardiac ejection fraction ≥50%; serum Cr ≤ 1.25 times normal range or creatinine clearance calculated by Cockcroft-Gault formula ≥45ml/min; ALT and AST≤ 3 times normal range, total bilirubin ≤ 1.5times normal range; （8）hemoglobin ≥ 80 g / L, neutrophils ≥ 1.0 × 10 ^ 9 / L, platelets ≥ 50 × 10 ^ 9 / L.

（9）INR≤ 1.5times normal range; APTT≤ 1.5times normal range; （10）Women in childbearing age must be not pregnant and do not plan pregnancy within 1 year of their cell transfusion; （11）Informed consent is signed by a subject or his lineal relation.

Exclusion Criteria:

1. Recent or current use of glucocorticoid or other immunosuppressor or Drug that stimulates bone marrow hematopoiesis;
2. Uncontrolled systemic active infection: fungi, bacteria, viruses or other infections;
3. Active infection with HBV, HCV or HIV;
4. Patients with symptoms and disease history of central nervous system;
5. Pregnant or lactating female；The patient did not agree to use effective contraception during the treatment period and for the following 1 year；
6. Patients receiving allogeneic hematopoietic stem cell transplantation, or organ transplantation
7. A history of other malignant tumors;
8. Primary immunodeficiency disease, or autoimmune disease;
9. Patients treated with PD-1 inhibitors or PD-L1 inhibitors prior to enrollment;
10. Patients who participated in other clinical trials within 4 weeks before blood collection;
11. Patients who had used CD19 targeted therapy before enrollment;
12. The investigator believes that there are other factors that are not suitable for inclusion or influence the subject's participation or completion of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of adverse events | 2 years
  Percentage of participants with adverse events

SECONDARY OUTCOMES:
objective remission rate | 3 months
  The percentage of participants who achieved complete remission (CR) and partial remission over all participants (ORR)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided